CLINICAL TRIAL: NCT00263159
Title: Pharmaceutical Care for Asthma Control Improvement
Brief Title: Pharmaceutical Care for Asthma Control Improvement (PHARMACI)-Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2005/320
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Pharmaceutical Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Pharmaceutical care for asthma patients

SUMMARY:
The objective of this study is to evaluate the therapeutic effectiveness and cost-effectivity of pharmaceutical care for asthma patients.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the therapeutic effectiveness and cost-effectivity of pharmaceutical care for asthma patients. Patients will be randomly allocated to the control group (= no input from pharmacist) or intervention group (= with pharmaceutical care at baseline and follow-up visits over 6 months).

ELIGIBILITY:
Inclusion Criteria:

* Patients with persistent asthma
* Asthma treatment for at least 12 months
* Regular visitors of the participating community pharmacy

Exclusion Criteria:

* Severe co-morbidity
* > 10 pack-years smoking history
* Asthma Control Test score < 15 or =25

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 221 (Actual)
Dates: Start 2006-01; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
The difference between study groups in the change of asthma control from baseline and follow-up visits | after 1, 3 and 6 months

SECONDARY OUTCOMES:
Peak flow | after 3 and 6 months
Knowledge of asthma and treatment | after 6 months
Asthma quality of life questionnaire (AQLQ) | after 6 months
Therapy adherence
Inhalation techniques | after 6 months
Smoking | after 6 months
Asthma exacerbations | after 6 months
General Practitioner (GP) visits, emergency room visits and hospitalisations
Working days lost and school days lost

CONTACTS AND LOCATIONS:
Overall Officials: Guy Brusselle, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Ghent — http://www.ugent.be